CLINICAL TRIAL: NCT07378917
Title: Evaluation of Metatarsophalangeal Joint Alignment in Mild and Moderate Hallux Abducto Valgus Through Orthotic Intervention
Brief Title: Orthotic Impact on MTP Alignment in Hallux Valgus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, CARMEN GARCÍA GOMARIZ, Associate Professor of Infirmary, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EJC_01
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hallux Valgus
Keywords: Hallux Abducto Valgus (HAV); Metatarsophalangeal Joint Alignment; Orthotic Devices; Radiographic Assessment
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthosis (Experimental): The study group will consist of 35 adult subjects, both men and women, diagnosed with mild to moderate Hallux Abducto Valgus (HAV) according to the Manchester scale.
  Interventions: Device: Hallux Valgus Orthosis

INTERVENTIONS:
Device: Hallux Valgus Orthosis — This study evaluates the effectiveness of an external hallux valgus orthosis in realigning the first metatarsophalangeal joint in patients with mild to moderate HAV. Two radiographic measurements of the valgus angle will be taken: at baseline and after 3 months of daily orthosis use. Participants will receive instructions for proper placement and adjustment. Secondary outcomes include pain (VAS), comfort, satisfaction, plantar pressure analysis (static/dynamic), device fit, and adherence. Data will be collected by podiatrists and anonymized for analysis.

SUMMARY:
This study aims to evaluate the effectiveness of an external corrector in realigning the first metatarsophalangeal joint in patients with mild to moderate Hallux Abducto Valgus, according to the Manchester scale. Changes in valgus angle will be assessed through radiographs, along with pain, comfort and adherence, comparing results with a control group.

DETAILED DESCRIPTION:
Introduction and Rationale Hallux Abducto Valgus (HAV) is the most common forefoot deformity, often associated with pain and functional limitations. Its development is multifactorial, and although surgical and conservative treatments exist, evidence regarding the real effectiveness of corrective orthopedic devices in early stages is scarce. This study seeks to provide scientific rigor to a device frequently recommended in clinical practice by evaluating its ability to correct alignment and improve symptoms.

Main and Secondary Objectives The primary objective is to assess the effectiveness of the corrector in realigning the first toe by measuring the valgus angle radiographically at three time points: without the corrector, immediately after application, and after 3 months. Secondary objectives include evaluating pain (VAS), comfort, adherence, device fit, changes in plantar pressure (static and dynamic), patient satisfaction, and differences compared to the control group.

Study Design and Population This is an experimental study involving a group of 35 subjects diagnosed with mild or moderate HAV according to the Manchester scale, recruited at the Aquilesia podiatry clinic (Vila-real, Castelló). Recruitment will be carried out through local media, social networks, and referrals from healthcare professionals. Informed consent, anonymity, and compliance with data protection regulations will be ensured.

Intervention and Measurements The intervention consists of applying an external hallux alignment corrector. Three radiographic measurements of the metatarsophalangeal angle will be taken: baseline, after corrector placement, and at 3 months. Additional data will include pain, comfort, adherence and device adjustment. Standardized scales (VAS, satisfaction questionnaires) and Excel-based data recording will be used.

Data Processing and Analysis Data will be collected by a podiatrist and anonymized before analysis. Intra- and intergroup differences will be evaluated using appropriate statistical tests, considering variables such as sex, age, and degree of deformity. The study aims to determine whether the corrector produces significant improvements in alignment and other clinical parameters, providing evidence for its usefulness in podiatric practice.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or female Age: 18 to 80 years Cooperative subject, informed of the need and duration of follow-up visits, ensuring full compliance with the protocol/study, and having signed informed consent No previous surgery on the foot and/or ankle Mild and/or moderate Hallux Valgus (Manchester Scale)

Exclusion Criteria:

* Patient with severe arteriopathy Patient with severe edema Patient with sensory neuropathy Patients who have used additional pharmacological treatments (analgesics/anti-inflammatories) during the entire study period Severe Hallux Valgus (Manchester Scale) Any systemic disease affecting the musculoskeletal system Rheumatoid arthritis involving the first metatarsophalangeal joint Instability of the first metatarsophalangeal joint History of previous foot and/or ankle surgery Hyperpronated foot with FPI >10 Severe pathological genu varum or valgum Pregnant women or suspected pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Valgus Angle Correction | 3 months
  Measurement of the hallux valgus angle on digital radiographs at baseline and after 3 months of orthosis use, to determine the degree of realignment of the first metatarsophalangeal joint.

SECONDARY OUTCOMES:
Pain Assessment (VAS) | 3 months
  Evaluation of pain intensity in the hallux region using the Visual Analog Scale (0 = no pain, 10 = worst pain).
Comfort and Satisfaction | 3 months
  Subjective assessment of comfort, aesthetics, and overall satisfaction with the orthosis through a structured questionnaire.
  Comfort was evaluated using a Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no comfort and 10 indicates maximum comfort.
Device Fit and Adjustment | 1day
  Evaluation of orthosis sizing and traction adjustment scored on a 1-10 scale, including ease of placement by the participant.
Orthosis Condition After Use | 3 months
  Assessment of wear and tear of the device after 3 months, scored on a 1-10 scale.
Adherence to Treatment | 3 months
  Monitoring of daily orthosis use through self-reported logs and follow-up visits.
Purchase Decision | 3 months
  Whether the participant would consider buying the orthosis after the study (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: CARMEN GARCÍA GOMARIZ, Principal Investigator — UNIVERSITAT DE VALÉNCIA DEPARTAMENTO D'INFERMERIA
Locations (1):
- Carmen García Gomariz, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No